CLINICAL TRIAL: NCT00610922
Title: RCT of Supplemented Docosahexaenoic Acid and Gross Motor Development Milestones in Healthy Infants.
Brief Title: Docosaexahenoic Acid and Gross Motor Milestones in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Prof. Carlo Agostoni, Dept of Pediatrics, San Paolo Hospital, University of Milan, Italy
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NEON-02/2005-DHA
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: Performance of motor skills
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental)
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) — DHA 20 mg per day through 12 months of life
  Arms: 2

SUMMARY:
To examine whether daily supplement of docosahexaenoic acid throughout the first year of life may speed up the achievement of gross motor development milestones in healthy infants, a total of 1160 healthy infants randomly allocated to receive throughout the first year of life daily oral supplement of vitamin D3 (400 IU) plus docosahexaenoic acid (20 mg) or vitamin D3 (400 IU) alone. Primary outcome measure: time of achieving gross motor development milestones. Secondary outcome measure: time of achieving early fine motor development milestones and language.

ELIGIBILITY:
Inclusion Criteria:

* weight at birth equal or above 2500 g;
* gestational age between 37 and 42 completed weeks;
* single birth;
* absence of neonatal or birth abnormalities;
* Apgar score greater than or equal to 7 at 5 m;
* white parents.

Exclusion Criteria:

* presence of neonatal diseases requiring hospitalisation for longer than 7 days;
* unknown father;
* parents unable to understand the protocol requirements and to fill out the infants diary;
* infant already enrolled or selected for another clinical study.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1160 (Actual)
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
time of achieving the four gross motor development milestones | 4, 8 and 12 months of age

SECONDARY OUTCOMES:
time of achieving early fine motor milestones and language | 4, 8 and 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Agostoni, Prof, Principal Investigator — Dept. of Pediatrics, San Paolo Hospital, University of MIlan, Italy

REFERENCES:
- [Derived] Agostoni C, Zuccotti GV, Radaelli G, Besana R, Podesta A, Sterpa A, Rottoli A, Riva E, Giovannini M. Docosahexaenoic acid supplementation and time at achievement of gross motor milestones in healthy infants: a randomized, prospective, double-blind, placebo-controlled trial. Am J Clin Nutr. 2009 Jan;89(1):64-70. doi: 10.3945/ajcn.2008.26590. Epub 2008 Dec 3. PMID 19056592